CLINICAL TRIAL: NCT05286931
Title: Evaluation of SpeeDx's Ciprofloxacin gyrA Assay for Clinical Care of STD Clinic Patients With Neisseria Gonorrhea
Brief Title: SpeeDx Ciprofloxacin gyrA Assay for N. Gonorrhoeae Gonococcal Infection
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Washington (Other)
Responsible Party: Principal Investigator, Lindley Barbee, Associate Professor: School of Medicine Allergy and Infectious Diseases, University of Washington
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: STUDY00012598
Record Dates: First submitted 2022-02-14; First posted 2022-03-18 (Actual); Last update posted 2022-03-18 (Actual); Status verified 2022-03

CONDITIONS: Neisseria Gonorrhoeae Infection
Keywords: antimicrobial resistance; ciprofloxacin; molecular diagnostics
MeSH Terms: conditions — Gonorrhea | interventions — Ciprofloxacin

STUDY DESIGN:
Intervention Model Description: Prospective cohort
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- N. gonorrhea (gyrA wildtype) -Ciprofloxacin Treatment Arm (Experimental): Participants who are N. gonorrhea (NG) positive and gyrA WT, will receive ciprofloxacin 500 mg PO x 1.
  Interventions: Drug: Ciprofloxacin 500 mg

INTERVENTIONS:
Drug: Ciprofloxacin 500 mg — Ciprofloxacin 500 MG, taken once orally.

SUMMARY:
This study aims to test the effectiveness of using of SpeeDx Resistance Plus assay to guide treatment of Neisseria gonorrhoeae (Ng) in a sexual health clinic setting.

DETAILED DESCRIPTION:
Patients entering the Sexual Health Clinic will be offered participation in the study if they have; 1) no infectious genitourinary symptoms that require immediate treatment, 2) who seek routine STI screening, 3) if they report sexual contact with a partner who reports having Ng or 4) men who have sex with men (MSM) with contact to chlamydia trachomatis (CT).

All participants will have specimen collected from anatomical sites of exposure for NAAT and culture. NAAT specimen positive for Ng will be flagged and further tested with SpeeDx Resistance Plus assay. This will delay results reporting on average by 1 day. The assay detects Ciprofloxacin resistance based on a point mutation of the gyrA gene (gyrA s91). Participants without this mutation or wild-type (gyrA WT) infection should be sensitive to Ciprofloxacin.

Participants who are N. gonorrhoeae (NG) positive and gyrA WT, will receive ciprofloxacin 500 mg PO x 1.

Participants with gyrA s91 mutation will be asked to return to clinic for the standard of care (i.e. ceftriaxone-based therapy).

ELIGIBILITY:
Inclusion Criteria:

* English speaking
* Have access to the internet (via computer or phone) on at least a weekly basis
* Asymptomatic (as defined below)

Exclusion Criteria:

* Urogenital symptoms consistent with a sexual transmitted infection (other than vaginitis associated with trichomonas vaginalis, bacterial vaginosis or yeast). Symptoms consistent with cervicitis, urethritis, or PID will not be offered enrollment.
* Antibiotic use within the last 2 weeks
* Contact to syphilis
* Contact to an STI and are unwilling to defer empiric treatment until diagnostic test results return
* Anyone receiving a gonococcal-active drug (such as Doxycycline, Penicillin, Ceftriaxone) during the visit. Those receiving metronidazole, fluconazole, or clotrimazole will not be excluded.
* Known allergy to ciprofloxacin and/or ceftriaxone

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 1800 (Estimated)
Dates: Start 2022-03-03 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Determine the number and proportion of Neisseria Gonorrhea (NG) cases that can be cured with ciprofloxacin | 2 years
  Number and proportion of patients who test positive for Neisseria Gonorrhea (NG) and are gyrA wildtype of all patients enrolled/screened for NG
To determine the effectiveness of treating patients with Neisseria Gonorrhea gyrA wildtype with Ciprofloxacin 500 mg orally once | 2 years
  Number and proportion of NG-positive patients with gyrA wildtype who are cured (i.e. have negative test of cure results) with 500mg ciprofloxacin overall and by anatomic site

SECONDARY OUTCOMES:
To confirm the SpeeDx gyrA Cipro-susceptibility prediction accuracy as compared to phenotypic susceptibility result | 2 years
  Percent concordance of gyrA result (molecular diagnostic) and the ciprofloxacin minimal inhibitory concentration (MIC) (aka. phenotypic antimicrobial susceptibility testing)
To determine time from screening to treatment using SpeeDx gyrA assay | 2 years
  Number of days between screening and treatment by treatment group (Ciprofloxacin or Standard of care)

CONTACTS AND LOCATIONS:
Overall Officials: Lindley Barbee, MD, MPH, Principal Investigator — University of Washington
Locations (1):
- Public Health -- Seattle & King County Sexual Health Clinic, Seattle, Washington, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Siedner MJ, Pandori M, Castro L, Barry P, Whittington WL, Liska S, Klausner JD. Real-time PCR assay for detection of quinolone-resistant Neisseria gonorrhoeae in urine samples. J Clin Microbiol. 2007 Apr;45(4):1250-4. doi: 10.1128/JCM.01909-06. Epub 2007 Jan 31. PMID 17267635
- [Background] Hooper DC, Wolfson JS. Fluoroquinolone antimicrobial agents. N Engl J Med. 1991 Feb 7;324(6):384-94. doi: 10.1056/NEJM199102073240606. No abstract available. PMID 1987461
- [Background] Allan-Blitz LT, Wang X, Klausner JD. Wild-Type Gyrase A Genotype of Neisseria gonorrhoeae Predicts In Vitro Susceptibility to Ciprofloxacin: A Systematic Review of the Literature and Meta-Analysis. Sex Transm Dis. 2017 May;44(5):261-265. doi: 10.1097/OLQ.0000000000000591. PMID 28407640
- [Background] Klausner JD, Bristow CC, Soge OO, Shahkolahi A, Waymer T, Bolan RK, Philip SS, Asbel LE, Taylor SN, Mena LA, Goldstein DA, Powell JA, Wierzbicki MR, Morris SR. Resistance-Guided Treatment of Gonorrhea: A Prospective Clinical Study. Clin Infect Dis. 2021 Jul 15;73(2):298-303. doi: 10.1093/cid/ciaa596. PMID 32766725
- [Background] Hadad R, Cole MJ, Ebeyan S, Jacobsson S, Tan LY, Golparian D, Erskine S, Day M, Whiley D, Unemo M; European collaborative group. Evaluation of the SpeeDx ResistancePlus(R) GC and SpeeDx GC 23S 2611 (beta) molecular assays for prediction of antimicrobial resistance/susceptibility to ciprofloxacin and azithromycin in Neisseria gonorrhoeae. J Antimicrob Chemother. 2021 Jan 1;76(1):84-90. doi: 10.1093/jac/dkaa381. PMID 32929456